CLINICAL TRIAL: NCT07176247
Title: Real-world Multicentre Study of AZtreonam-AVIbactam Treatment With Infections or Suspected Infections Caused by Multidrug-resistant Gram-negative Bacteria
Acronym: AZAVI
Status: Enrolling by invitation | Type: Observational
Sponsor: French Society for Intensive Care (Other)
Collaborators: SPILF (Unknown)
Responsible Party: Sponsor
Other Study IDs: CE-SRLF 25-034
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Critical Care; Infection; Antibiotic Resistance; Infectious Diseases
Keywords: aztreonam; avibactam; critical care; infectiology; antibiotic; resistance; new betalactam; aztreonam-avibactam; real-world
MeSH Terms: conditions — Infections; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized patients under Aztreonam-Avibactam
  Interventions: Drug: Aztreonam-Avibactam

INTERVENTIONS:
Drug: Aztreonam-Avibactam — Antibiotic therapy with Aztreonam-Avibactam

SUMMARY:
The AZAVI study is a multicenter observational registry (ICU and Infectious Diseases departments), designed to evaluate the real-world use of aztreonam-avibactam for suspected or documented infections caused by metallo-β-lactamase (MBL)-producing Enterobacterales or highly resistant Gram-negative bacteria. The study combines a retrospective cohort (patients treated during the 12 months prior to the drug's hospital availability) and a prospective cohort (patients consecutively included over 24 months).

The primary outcome is clinical success at day 7 after antibiotic discontinuation, defined as resolution of signs and symptoms of infection without recurrence or need for additional active therapy. Secondary outcomes include microbiological eradication, 14-day and 28-day all-cause mortality, infection relapse, length of stay, safety outcomes, and predictors of treatment failure.

Data will be collected using a standardized CRF, including demographics, severity scores, infection site and pathogens, therapeutic regimens, organ failures and support, adverse events, and outcomes. Descriptive statistics and multivariable models will be used to assess real-world effectiveness, identify determinants of clinical response, and inform stewardship strategies. This registry will provide the first national-scale evidence on the role of aztreonam-avibactam in critically ill patients outside the framework of controlled clinical trials.

DETAILED DESCRIPTION:
1. Background and Rationale The emergence of carbapenemase-producing bacteria, particularly metallo-β-lactamase (MBL) producers such as NDM, poses a major therapeutic challenge in intensive care settings. Current guidelines recommend combining ceftazidime-avibactam (CAZ-AVI) with aztreonam for these infections, but these were developed before the availability of the fixed combination aztreonam-avibactam (ATM-AVI). ATM-AVI offers a more targeted option by pairing a β-lactam stable to MBL hydrolysis with a non-metallo β-lactamase inhibitor. While in vitro and limited in vivo data are promising, real-world evidence remains scarce.
2. Objectives

   -Primary Objective: To describe the frequency of clinical success of ATM-AVI in patients treated for suspected or documented MBL-producing bacterial infections.

   -Secondary Objectives: To assess microbiological and clinical effectiveness. To describe the emergence of resistance during treatment. To identify predictors of clinical and microbiological response. To evaluate ICU and hospital length of stay, mechanical ventilation duration, and all-cause mortality at day 28 and day 90.

   To assess safety and adverse events. To compare prescribing practices between infectious diseases and intensive care units.
3. Study Design

   Multicenter, observational study with both retrospective and prospective cohorts:
   * Retrospective arm: Patients treated with ATM-AVI in the 12 months preceding study initiation.
   * Prospective arm: Patients treated with ATM-AVI over a 24-month period following study initiation.

   Participating centers include ICUs and infectious diseases departments recruited via national professional networks.
4. Population

   * Inclusion criteria: Hospitalized patients with suspected or documented infection due to MBL-producing bacteria, treated with ATM-AVI.
   * Exclusion criteria: Explicit refusal by patient or legal representative.
5. Endpoints

   -Primary endpoint: Clinical success at the test-of-cure visit, day 7 after completion of the initial ATM-AVI regimen, defined as resolution of infection signs and symptoms without need for further active antibiotics. Death (any cause) and microbiologically confirmed relapse are considered treatment failures.

   -Secondary endpoints: Microbiological eradication/persistence. Mortality at day 28 and day 90. Duration of hospitalization, ICU stay, and mechanical ventilation. Adverse events attributable to ATM-AVI. Patterns of monotherapy vs. combination therapy.
6. Data Collection

   * Retrospective arm: Identification of cases via ICD-10 coding (infections due to multidrug-resistant organisms), microbiology laboratory records (MBL-positive isolates), pharmacy dispensing data, and early access registries.
   * Prospective arm: Data collected at the time of ATM-AVI prescription and during follow-up.

   All data are pseudonymized and entered into a secure electronic case report form.
7. Statistical Analysis Descriptive statistics for baseline characteristics and outcomes. Univariate and multivariate analyses to identify predictors of clinical success at day 7 post-treatment.

Propensity score analysis to compare monotherapy vs. combination therapy. All tests two-sided, p < 0.05 considered significant. Expected Results and Impact

In total, This study will provide real-world data on the effectiveness, safety, and resistance dynamics of ATM-AVI in severe infections due to MBL-producing bacteria. Results will support clinical decision-making and help refine treatment strategies in critical care and infectious diseases settings.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with suspected or documented infection due to MBL-producing bacteria, treated with ATM-AVI.

Exclusion Criteria:

* Explicit refusal by patient or legal representative.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients with suspected or documented infection due to MBL-producing bacteria, treated with ATM-AVI.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical success at the test-of-cure visit (day 7 after completion of initial antibiotic therapy) | day 7 after completion of initial antibiotic therapy
  Clinical success at the test-of-cure visit, day 7 after completion of the initial ATM-AVI regimen, defined as resolution of infection signs and symptoms without need for further active antibiotics. Death (any cause) and microbiologically confirmed relapse are considered treatment failures.

SECONDARY OUTCOMES:
Microbiological eradication/persistence | Day-28
Mortality | Mortality at day 28 and day 90
Duration | Day-28
  Duration of hospitalization, ICU stay, and mechanical ventilation
Adverse events attributable to ATM-AVI | Day-28
Patterns of monotherapy vs. combination therapy | Day-28

CONTACTS AND LOCATIONS:
Locations (1):
- French Society of Intensive Care (SRLF), Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Access Criteria: The datasets generated during and/or analyzed during the study are available from the corresponding author on reasonable request.